CLINICAL TRIAL: NCT03303014
Title: Use of 5-0 Prolene Versus 5-0 Fast Absorbing Gut During Cutaneous Wound Closure: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: 5-0 Prolene Versus 5-0 Fast Absorbing Gut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 811023; NCT02991755 (obsolete NCT alias)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Cutaneous Wound
Keywords: Suture; Absorbable; Non-absorbable; Split wound; Cutaneous Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-0 Prolene (Experimental): Half of the wound will be treated with 5-0 prolene
  Interventions: Device: 5-0 Prolene, 5-0 Fast Absorbing Gut
- 5-0 Fast Absorbing Gut (Experimental): Half of the wound will be treated with 5-0 fast absorbing gut
  Interventions: Device: 5-0 Prolene, 5-0 Fast Absorbing Gut

INTERVENTIONS:
Device: 5-0 Prolene, 5-0 Fast Absorbing Gut — The interventions are two types of sutures: 5-0 Prolene, 5-0 Fast Absorbing Gut.

SUMMARY:
When using suture (stitches) to close wounds, surgeons can use suture that is absorbable or non-absorbable. Absorbable sutures naturally break down. Non-absorbable sutures need to be removed. We wish to determine how the cosmetic result of a specific absorbable suture (fast absorbing gut) compares to that of a specific non-absorbable suture (prolene).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of 5-0 prolene during repair of linear cutaneous surgery wounds improves scar cosmesis compared to wound closure with 5-0 fast absorbing gut (both SOC). We will use a split wound model, where half of the wound is treated with 5-0 prolene and the other half is repaired with 5-0 fast absorbing gut. Three-months post-surgery, the scar will be measured via the physician observer scar assessment scale, a validated scar instrument (research procedure). The scar width and adverse events will be recorded.

There are many options when it comes to closing a linear cutaneous wound, and an important consideration is choosing between non-absorbable and absorbable sutures. The overall aesthetic superiority between the two is not well understood. Studies to date have typically compared prolene (non-absorbable) and vicryl (absorbable) sutures and found no significant difference in cosmesis.1-4 One study found an increased pain score at 10 days with vicryl, but not at 6 weeks,1 while others have found no difference in pain.2-4 Another study found an increased number of complications with vicryl sutures, including infections and suture granulomas.4 This supports past observations that absorbable sutures can cause more of an immune response and therefore inflammation, despite the benefit of providing more prolonged support to wound edges compared to non-absorbable sutures.1

There is a lack of data, though, comparing prolene to other absorbable sutures, such as fast absorbing gut. In the setting of blepharoplasty, a study found that a running stitch of fast absorbing gut with a simple interrupted stitch of prolene at each end of the incision yielded better cosmetic results and fewer complications than a running stitch or subcuticular stitch using prolene.5 More studies are therefore needed to compare the outcomes of linear closures using only prolene compared to only fast absorbing gut. Using only absorbable sutures has the potential benefit of decreasing healthcare costs by reducing the number of appointments needed for suture removals, and, if superior in terms of cosmesis, corrective procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head and neck with predicted primary closure
* Willing to return for follow up visit.

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale (POSAS) | within 3 months of the procedure
  The primary endpoint will be the score of two blinded reviewers using the physician observer assessment score at a three-month assessment visit.

SECONDARY OUTCOMES:
Width of the scar | within 3 months of the procedure
  The secondary endpoint will include the width of the scar at the follow-up visit and any complications from the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zemla J. [Plastic operation of the alveolar process and associated deformities of the middle part of the face after primary operations for bilateral complete clefts of the lip, alveolar process and palate]. Protet Stomatol. 1977 Mar-Apr;27(2):143-4. No abstract available. Polish. PMID 270137
- [Background] Erel E, Pleasance PI, Ahmed O, Hart NB. Absorbable versus non-absorbable suture in carpal tunnel decompression. J Hand Surg Br. 2001 Apr;26(2):157-8. doi: 10.1054/jhsb.2000.0545. PMID 11281671
- [Background] Theopold C, Potter S, Dempsey M, O'Shaughnessy M. A randomised controlled trial of absorbable versus non-absorbable sutures for skin closure after open carpal tunnel release. J Hand Surg Eur Vol. 2012 May;37(4):350-3. doi: 10.1177/1753193411422334. Epub 2011 Oct 10. PMID 21987279
- [Background] Menovsky T, Bartels RH, van Lindert EL, Grotenhuis JA. Skin closure in carpal tunnel surgery: a prospective comparative study between nylon, polyglactin 910 and stainless steel sutures. Hand Surg. 2004 Jul;9(1):35-8. doi: 10.1142/s0218810404002017. PMID 15368623
- [Background] Joshi AS, Janjanin S, Tanna N, Geist C, Lindsey WH. Does suture material and technique really matter? Lessons learned from 800 consecutive blepharoplasties. Laryngoscope. 2007 Jun;117(6):981-4. doi: 10.1097/MLG.0b013e31804f54bd. PMID 17545862